CLINICAL TRIAL: NCT05133427
Title: High-Intensity Focused Ultrasound (HIFU) for Treatment of Non-nodular and Recurrent Basal Cell Carcinomas of the Skin: Efficacy and Safety.
Brief Title: HIFU for Treatment of Non-nodular and Recurrent BCC
Acronym: BCC-HIFU2101
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joergen Serup (Other)
Collaborators: Zealand University Hospital (Other)
Responsible Party: Sponsor-Investigator, Joergen Serup, Professor, Chief Physician, Department of Dermatology, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIV-21-06-037051
Record Dates: First submitted 2021-10-29; First posted 2021-11-24 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Basal Cell
Keywords: Basal cell carcinoma; BCC; Skin cancer; High intensity focused ultrasound; HIFU; Dermatology
MeSH Terms: conditions — Carcinoma, Basal Cell; Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: The study is a multicenter (two-center), open-label study in humans (hospital outpatients). The study is not comparative with respect to the two study groups; however, it is aimed to pool data if the study groups are statistically comparable.
  The investigation is performed prior to CE mark to confirm safety and performance of the System ONE-M device when used as intended, i.e. as an non-invasive method to remove non-nodular basal cell carcinoma by 20 MHz high intensity focused ultrasound.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Areas with de-novo or recurrent BCC (Experimental): Areas with non-nodular de-novo or recurrent BCC area will be treated by high intensity focused ultrasound.
  Interventions: Device: TOOsonix system ONE-M

INTERVENTIONS:
Device: TOOsonix system ONE-M — All selected BCC areas will be treated by high intensity focused ultrasound

SUMMARY:
The overall objective of this study is to demonstrate the safety and efficacy of removal of Basal Cell Carcinoma (BCC) using a new investigational equipment based on high-intensity focused ultrasound.

Basal cell carcinoma is the most common cancer in Europe, Australia and the U.S.A. The general upwards age shift in the population in these regions is expected to be accompanied by an increase in the incidence of this type of cancer. There are currently more the 20.000 BCC registrations in Denmark every year, and occurrences on a global scale are counted in several tens of millions per year. Finding new and more effective treatment methods are therefore highly relevant from both a clinical and socioeconomic perspective.

The investigational device used in the investigation is a Danish developed system capable of making controlled and targeted thermo-mechanical treatment of small intradermal volumes containing e.g. BCC cells, but without inflicting damage to the surrounding tissue.

The investigation involves an evaluation of the safety and efficacy profile 3 months after a single 3-5 minute treatment. Subsequent follow-up of secondary endpoints is done every third month until the end of the study one year after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of each gender aged 18 years or older at the time of informed consent. There is no upper limit of age.
* Subjects who have received oral and written study information, accepted participation and signed the informed consent document.
* Subjects who are willing and mentally and physically capable to understand and follow the treatment and follow-up schedule including post-treatment care instructions.
* Subjects who are willing to have photographs and images taken of the treated lesions to be used anonymously or coded in evaluations and publications.
* Subjects, who have histologically and clinically verified basal cell carcinoma either as newly diagnosed non-nodular cancer (one group) or as a recurrent cancer in a local site (another group) previously treated with any method practiced in dermatology clinics, hospital or the primary sector. Tumors of thickness more than 2.0 mm measured by ultrasound or OTC are considered of the "nodular" type. Thus, only tumors of thickness 2.0mm and less are included.

Exclusion Criteria:

* Subjects who are less than 18 years at the time of informed consent.
* Subject is pregnant or lactating at time of first treatment
* Subjects with extensive, invasive or advanced skin cancer when another method in use such as radiotherapy or Mohs' surgery has priority and offers the patient better opportunity of cure.
* Cancers on anatomical sites where the ultrasound probe cannot be adapted for anatomical reasons
* Any systemic disease that according to investigator's assessment may interfere with the spontaneous course of a skin cancer.
* Any condition predisposing to treatment-related adverse effects or complications from the ultrasound treatment.
* Subjects with abnormal scar formation
* Subjects with impaired wound healing
* Subjects with the basal cell carcinoma under study located nearby (<5 cm) an implant or a site injected with a dermal filler or paraffin.
* Subjects with any other acute or chronic condition which, in the opinion of the investigator, could interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Cure Rate | 3 months
  Cure rate of basal cell carcinoma (de novo or recurrences after conventional treatments, two groups) following treatment with the investigational device. Measured as a binary Yes/No output.
Severity of short term treatment side effects | 3 months
  Safety profile after treatment of basal cell carcinoma (de novo or recurrences after conventional treatments, two groups) following treatment with the investigational device. Measured on a 4-point severity score ranging from No side effects (score 1) to Severe side effects (score 4).

SECONDARY OUTCOMES:
Severity of adverse events | 12 months
  Any objective adverse effect or event, local or systemic, related to the treatment and the investigational device (wound and course of wound healing, scar formation, instrumental hazards) measured at 6, 9 and 12 months. Measured on a 4-point severity score ranging from No side effects (score 1) to Severe side effects (score 4).
Cure Rate | 12 months
  Cure rate of basal cell carcinoma (de novo or recurrences after conventional treatments, two groups) following treatment with the investigational device measured at 6, 9 and 12 months. Measured as a binary Yes/No output.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen, Capital Region
  - Roskilde Hospital, Roskilde, Region Sjælland

IPD SHARING:
Plan to Share IPD: No